CLINICAL TRIAL: NCT06881927
Title: Reduction in ImmunoSuppressive Regimen Among Kidney Transplant Recipients Patients Admitted to the Intensive Care Unit for Septic Shock and/or Acute Respiratory Failure: a Multicenter, Open-label, Phase IIb Randomized Controlled Trial
Brief Title: Eduction in ImmunoSuppressive Regimen Among Kidney Transplant Recipients Patients Admitted to the Intensive Care Unit for Septic Shock and/or Acute Respiratory Failure
Acronym: REDIS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9416
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-03

CONDITIONS: Sepsis and Septic Shock; Acute Respiratory Failure; Kidney Transplant Recipients; Immunosuppressive Agents
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — hydrocortisone hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reduction of the level of immunosuppression (Experimental): In this arm, the usual immunosuppressive treatment of the patients will be discontinued.
  Patients will receive hydrocortisone hemisuccinate 200 mg per day (slow direct intraveinous injection of 50 mg four times a day, or through an electric syringe pump).
  Interventions: Other: reduction of the level of immunosuppression
- usual immunosuppression maintenance (Active Comparator): In this group: patients will receive hydrocortisone hemisuccinate 200 mg per day (slow direct intraveinous injection of 50 mg four times a day, or through an electric syringe pump).
  The usual treatment with immunosuppressive agents will be continue: calcineurin inhibitors and/or mTOR inhibitors and/or Azathioprine, and/or Mycophénolate Mofétil (MMF)/Mycophenolice Acide (MPA).
  For MMF/MPA, at the discretion of the treating clinicians, dosage may be reduced or drug discontinued.
  Interventions: Drug: Hydrocortisone Hemisuccinate: 200 mg per day.

INTERVENTIONS:
Drug: Hydrocortisone Hemisuccinate: 200 mg per day. — The hydrocortisone hemisuccinate is a powder and solvent for injectable solution at 100 mg. The powder must be dissolved in the solvent to ensure final isotonicity. The solution must be used within 24 hours. The injection is performed as a slow direct IV injection, either via an electric syringe pump or as a bolus of 50 mg every 6 hours
  Arms: usual immunosuppression maintenance
Other: reduction of the level of immunosuppression — In this arm, the usual immunosuppressive treatment of the patients will be discontinued.
  Patients will receive hydrocortisone hemisuccinate 200 mg per day (slow direct intraveinous injection of 50 mg four times a day, or through an electric syringe pump).
  Arms: reduction of the level of immunosuppression

SUMMARY:
Kidney transplantation is the treatment of choice for end-stage chronic kidney disease. Kidney transplantation is at the first rank of solid organ transplantation in France, with 3,376 grafts performed in 2022. Immunosuppressive therapy, required to prevent graft rejection, exposes graft recipients to complications related to decreased immunity, including opportunistic infections and neoplastic complications.

After the earlt post-transplantation period, up to 10% of kidney transplant recipients will require admission to the intensive care unit (ICU). The main reasons for admission are septic shock and acute hypoxemic respiratory failure. ICU stay has a significant impact on these patients with a mortality rate reaching 40%, that remains increased even after ICU discharge. Furthermore, an impact on graft function has been demonstrated, with deterioration of graft function in 1/3 of patients, and among those, up to one in two will require resumption of renal replacement therapy (RRT).

Although the occurrence of septic shock or acute respiratory failure related to an infection is more common and severe, the optimal management strategy for immunosuppressors is not defined in kidney transplant recipients admitted to the ICU in those settings.

Maintain a high level of immunosuppressive therapies may hinder the recovery from the acute critical condition. Furthermore, these treatments have a narrow therapeutic index; for instance, the management of calcineurin inhibitors is challenging in the ICU due to pharmacodynamic changes associated with the acute situation (distribution volume, organ failure) and the numerous potential drug interactions that carry inherent risks of overdose.

the investigators hypothesize that a reduction in the level of immunosuppressive treatments could promote recovery in kidney transplant recipients admitted to the ICU for septic shock and/or acute hypoxemic respiratory failure, without adversely affecting the risk of rejection or long-term renal prognosis.

ELIGIBILITY:
Inclusion Criteria:

* - Adult patients, aged 18 years-old and over,
* Kidney transplant recipients, with transplantation occurring more than 3 months prior to ICU admission
* Patients admitted to the ICU in the setting of:

  * Septic shock (sepsis requiring vasopressor support, with or without hyperlactatemia),
  * And/or acute respiratory failure of presumed infectious origin (invasive or non-invasive ventilation, FiO2 greater than or equal to 50%),
* Patients treated with at least an immunosuppressive bitherapy (including steroids, calcineurin inhibitors, mTOR inhibitors, azathioprine, or mycophenolate mofetil),
* Patients affiliated with a social health insurance protection scheme,
* Patients able of understanding the objectives and risks related to the research and providing a dated and signed informed consent. If patient is unable to consent: consent from relatives will be searched, and if absent, an emergency procedure will be process.
* Women of childbearing potential, provided they have a negative blood pregnancy test on the day of the inclusion visit.

Exclusion Criteria:

* Minor patients,
* Patients unable to consent: under legal protection measures, patients deprived of liberty,
* Kidney transplant recipients treated with Belatacept due to the persistent effect of Belatacept, it is not possible to modulate this treatment in a short term period,
* Patients with severe chronic graft dysfunction (glomerular filtration rate < 20 ml/min/1.73m² according to the CKD-EPI formula in the month prior to admission),
* Transplant renal recipients who have already resumed RRT (hemodialysis or peritoneal dialysis),
* Multi-organ transplant recipients,
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the rate of patients showing a change in the SOFA (Sequential Organ Failure Assessment) score of at least 4 points | Day 5
  SOFA score is a usual score used to assess gravity and its evolution among critically ill patients (ICM 1996)

IPD SHARING:
Plan to Share IPD: No